CLINICAL TRIAL: NCT03530085
Title: Decitabine+ Fludarabine+Busulfan Conditioning Regimen for Elderly Acute Myeloid Leukemia in Complete Remission Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Dec+Flu+Bu Conditioning Regimen for Elderly AML in CR Undergoing Allo-HSCT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Guangzhou First People's Hospital (Other); Peking University People's Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dec+FB-Elderly AML-2018
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Acute Myeloid Leukemia; Allogeneic Hematopoietic Stem Cell Transplantation; Conditioning; Elderly
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Busulfan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dec+Flu+Bu Conditioning Regimen (Experimental): For AML patients older than 60 years in CR, Decitabine+ Fludarabine+Busulfan conditioning regimen was used (Decitabine 20mg/m2/day on days -9 to -7；Fludarabine(Flu) 30mg/m2/day on days -6 to -3；Busulfan (BU) 3.2 mg/kg/day on days -5 to -4).
  Interventions: Drug: Decitabine; Drug: Busulfan (BU); Drug: Fludarabine(Flu)

INTERVENTIONS:
Drug: Decitabine — Decitabine was administered at 20mg/m2/day on days -9 to -7.
Drug: Busulfan (BU) — Busulfan was administered at 3.2 mg/kg/day on days -5 to -4.
Drug: Fludarabine(Flu) — Fludarabine(Flu) was administered at 30mg/m2/day on days -6 to -3.

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is reported to be able to improve the outcomes for elderly acute myeloid leukemia (AML) in complete remission (CR). At present, the best conditioning regimen for elderly AML in CR remains in discussion. In this prospective study, the safety and efficacy of Dec+Flu+Bu myeloablative conditioning regimens in patients with elderly AML in CR undergoing allo-HSCT are evaluated.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is reported to be able to improve the outcomes for elderly AML(older than 60 years) in complete remission (CR). At present, the best conditioning regimen for elderly AML in CR remains in discussion. Flu+Bu conditioning regimen is the most commonly used regimen for elderly AML in CR undergoing allo-HSCT. However, it appears to have higher relapse rate. To reduce the relapse rate, decitabine is added in the conditioning regimen. In this prospective study, the safety and efficacy of Decitabine+ Fludarabine+Busulfan myeloablative conditioning regimens in patients with elderly AML in CR undergoing allo-HSCT are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* AML patients older than 60 years, younger than 80 years
* In complete remission before transplantation
* With HLA-matched sibling donors

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | 2 year

SECONDARY OUTCOMES:
disease-free survival (DFS) | 2 year
relapse | 2 year
transplant-related mortality (TRM) | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Department of Hematology,Nanfang Hospital
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Q, Hu Z, Xu N, Jiang Y, Fan Z, Huang F, Lin R, Jin H, Zeng Y, He H, Zhu P, Yu G, Shi P, Sun R, Xu X, Li Z, Zhang Y, Sun J, Wang Y, Xuan L. Decitabine combined with reduced-intensity conditioning for older patients with acute myeloid leukemia in composite complete remission undergoing allogeneic hematopoietic stem cell transplantation: a multicenter, single-arm, phase 2 trial. Lancet Reg Health West Pac. 2025 Aug 12;61:101664. doi: 10.1016/j.lanwpc.2025.101664. eCollection 2025 Aug. PMID 40831735